CLINICAL TRIAL: NCT07049224
Title: The Effectiveness of a Diet With Beef as Key Protein Component Versus a Plant-Based Diet to Support Integrated Muscle Protein Synthesis Rates in Healthy Older Individuals
Acronym: OmniVeg_Diet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 24-025; NL87069.068.24 (Other: Toetsing Online)
Record Dates: First submitted 2024-12-19; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-12

CONDITIONS: Muscle Protein Synthetic Response to Protein
MeSH Terms: interventions — Diet, Western; Diet, Plant-Based; Diet, Vegan

STUDY DESIGN:
Intervention Model Description: Randomized, counter-balanced, cross-over design, researchers and participants are not blinded, analysts are blinded.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEAT-PLANT (Experimental): Participants will be subjected to a 10-day diet containing meat and animal products, followed by a 10-day diet containing plant products. During the interventional period participants will perform unilateral lower limb resistance exercise.
  Interventions: Other: Meat diet; Other: Plant diet
- PLANT-MEAT (Experimental): Participants will be subjected to a 10-day diet containing plant products, followed by a 10-day diet containing meat and animal products. During the interventional period participants will perform unilateral lower limb resistance exercise.
  Interventions: Other: Meat diet; Other: Plant diet

INTERVENTIONS:
Other: Meat diet — Participants will be subjected to a 10-day diet containing meat and animal products. During the interventional period participants will perform unilateral lower limb resistance exercise.
  Other Names: Omnivorous diet
Other: Plant diet — Participants will be subjected to a 10-day diet containing plant products. During the interventional period participants will perform unilateral lower limb resistance exercise.
  Other Names: Vegan diet

SUMMARY:
Muscles are composed out of proteins. These proteins in turn are composed out of smaller building blocks, called amino acids. By consuming a sufficient amount of dietary protein, a sufficient amount of amino acids become available to build new muscle proteins. The body's ability to build these new muscle proteins is of great importance to maintain muscle strength and function.

Previous research suggests that a meal containing proteins from meat results in a better stimulation of the body's ability to build muscle proteins, when compared to a meal containing only plant-based proteins. However, these previous studies have only been performed following the ingestion of a single meal. As a result it is currently unknown how the muscles respond to a more prolonged ingestion of a diet containing animal/meat products, in comparison to a plant-based diet. Therefore, this study aims to investigate how fast new muscle proteins are being build when consuming a diet containing animal/meat products, in comparison to a plant-based (vegan) diet.

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex
* Aged between 65 and 85 y inclusive
* BMI between 18.5 and 30 kg/m2 inclusive

Exclusion Criteria:

* Not willing to consume meat/animal-based products during the study period
* Any food allergies (e.g. milk, gluten, etc.)
* Participating currently or in the 3 months prior to the study in a structured progressive exercise program.
* Smoking
* History of cardiovascular, respiratory, gastrointestinal, urogenital, neurological, psychiatric, dermatologic, musculoskeletal, metabolic, endocrine, haematological, immunologic disorders, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol, interfere with the execution of the experiment, or potential influence the study outcomes (to be decided by the study team and responsible physician)
* Diagnosed with phenylketonuria (PKU)
* Donated full blood 3 months prior to test day
* Use of any medications that interferes with study participation and/or outcomes (i.e. corticosteroids, non-steroidal anti-inflammatories, gastric acid suppressing medication) as assessed by the study team and responsible medical doctor.
* Use of DOAC, vitamin-K-antagonist, or multiple anticoagulants
* Fasting blood glucose >7 mmol/L

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Healthy older males and females are eligible to participate
Enrollment: 32 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Integrated muscle protein synthesis rate in rested leg | The 2 intervention periods over which FSR is determined will each last 10 days
  The main study endpoint will be the difference in muscle protein synthesis rates in the non-exercised leg, between the plant-based diet and the meat diet, expressed as FSR (%/day).

SECONDARY OUTCOMES:
Integrated muscle protein synthesis rate in exercised leg | The 2 intervention periods over which FSR is determined will each last 10 days
  The difference in muscle protein synthesis rates in the exercised leg, between the plant-based diet and the meat diet, expressed as FSR (%/day).
Blood glucose | The 2 intervention periods after which the outcomes are determined will each last 10 days
  The difference in plasma glucose concentrations will be determined following the MEAT vs PLANT diet
Blood insulin | The 2 intervention periods after which the outcomes are determined will each last 10 days
  The difference in plasma, insulin, will be determined following the MEAT vs PLANT diet
Blood lipid profile | The 2 intervention periods after which the outcomes are determined will each last 10 days
  The difference in blood lipid profile will be determined following the MEAT vs PLANT diet
Blood inflammatory markers | The 2 intervention periods after which the outcomes are determined will each last 10 days
  The difference in blood inflammatory markers will be determined following the MEAT vs PLANT diet
Blood amino acid profile | The 2 intervention periods after which the outcomes are determined will each last 10 days
  The difference in plasma amino acid profile will be determined following the MEAT vs PLANT diet
Blood pressure | The 2 intervention periods after which the blood pressure is determined will each last 10 days
  The difference in blood pressure (both systolic and diastolic) will be determined following the MEAT vs PLANT diet

OTHER OUTCOMES:
Participant characteristics | At baseline, before start interventional period
  Participants characteristics at baseline will be reported as descriptives. This includes: Age, sex, body mass, height, BMI, Body composition as assed by DEXA scan, habitual dietary intake, habitual physical activity.
Muscle histology characteristics | At baseline, before start interventional period
  Muscle histology characteristics at baseline will be reported as descriptive.
Muscle signaling proteins | The 2 intervention periods over which muscle signaling proteins are determined will each last 10 days
  The difference in muscle signaling protein between the plant-based diet and the meat diet.
Dietary intake | The 2 intervention periods that will be compared will each last 10 days
  The dietary intake during the 2 interventional periods will be compared. Measured by dietary intake records
Fecal Microbiome | The 2 intervention periods that will be compared will each last 10 days
  The Fecal microbiome following the 2 interventional periods will be compared, measured in fecal samples
Step count | The 2 intervention periods that will be compared will each last 10 days
  The step count during the 2 interventional periods will be compared. Measured by an Actigraph activity monitor
Subjective feeling | The 2 intervention periods that will be compared will each last 10 days
  Satiety, muscle soreness, and gastro-intestinal complaints scores during the 2 interventional periods will be compared. Measured by visual analog scale questionnaires. The left side of the 100mm scale represents a score of 0 (= no complaints). The right side of the 100mm scale represents a score of 100 (=severe complaints)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided